CLINICAL TRIAL: NCT06990243
Title: Reliability and Validity of the Turkish Version of the Spinal Cord Injury Pain Instrument
Brief Title: Reliability and Validity of the Turkish Version of the SCIPI
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Lecturer, Istinye University
Other Study IDs: 15
Record Dates: First submitted 2025-04-19; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Neuropathic Pain; Spinal Cord Injury
Keywords: Neuropathic pain; Psychometric properties; Spinal cord injury pain instrument
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation Group — An evaluation form will record the participants' socio-demographic characteristics and information about their disease/treatment. Consciousness and cognitive tests will be performed. Then, pain will be assessed with the Visual Analog Scale, 4-Question Neuropathic Pain Questionnaire,, and the Spinal Cord Injury Pain Instrument (SCIPI).

SUMMARY:
Pain after spinal cord injury (SCI) is common, with the majority of individuals experiencing chronic pain and a significant portion reporting severe pain that interferes with their daily lives. Pain due to SCI is divided into two main groups: nociceptive and neuropathic. Clinical expertise is required for the accurate classification of these types of pain. Existing screening tools are generally evaluated with heterogeneous samples and therefore have limited accuracy in individuals with SCI. To address this deficiency, the Spinal Cord Injury Pain Instrument (SCIPI) was developed to define neuropathic pain in a manner specific to SCI. The SCIPI consists of seven items that assess the characteristics of pain and triggering factors. Although this scale, developed in English, has been translated into different languages, there is no Turkish version. This study aimed to examine the validity and reliability of the Turkish version of the SCIPI.

DETAILED DESCRIPTION:
Pain after spinal cord injury (SCI) is a common problem. Approximately 80% of individuals with SCI experience chronic pain, while one-third experience pain severe enough to interfere with their daily lives. Pain in individuals with SCI is divided into two main categories: nociceptive pain and neuropathic pain. Nociceptive pain is defined as pain that occurs when sensory receptors in peripheral nerves detect and encode noxious stimuli, while neuropathic pain is defined as pain that occurs as a result of a lesion or disease of the somatosensory nervous system. The classification of pain types is made both by the spinal cord injury pain classification developed by the International Association for the Study of Pain (IASP) and its successors. However, clinical expertise is required to apply these classifications correctly. For this reason, various screening tools have been developed over the years to more easily distinguish between neuropathic pain and non-neuropathic pain. These tools are usually based on a combination of physical examination findings and self-report or on self-report alone. However, existing tools have generally been evaluated with samples with heterogeneous etiologies and have been found to have lower accuracy rates in individuals with spinal cord injury.

In response to the need for a screening tool that is both sensitive and specific to distinguish neuropathic pain in individuals with SCI, the Spinal Cord Injury Pain Scale (SCIAS) was developed. This tool consists of seven features developed in light of clinical experience and literature analysis to distinguish neuropathic pain. These features include pain descriptions, pain triggered by dynamic touch, factors that increase and decrease pain, timing of pain, and pain felt in sensitive areas. Although the SCIAS has similar features to other pain screening tools, it has the potential to better distinguish the specific nature of pain associated with SCI.

The SCIAS, which was developed in English, has been translated into Chinese, French, and Portuguese. A Turkish version is needed. This study aimed to examine the reliability and validity of the Turkish version of the SCIAS.

ELIGIBILITY:
Inclusion Criteria:

* Having any level of SCI
* Being 18-70 years old
* Being at least one month since the SCI
* Being inpatient rehabilitation or living in the community

Exclusion Criteria:

* Having major depression
* Having suicidal intent or plans
* Being currently addicted to alcohol or drugs
* Not taking stable doses of psychoactive medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with spinal cord injuries
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
The Spinal Cord Injury Pain Instrument (SCIPI) | 1 week
  SCIPI was developed by Dr. Martin B. Forchheimer et al. to screen for neuropathic pain after spinal cord injury. It is an interview-based assessment tool designed to screen for neuropathic pain in individuals with SCI. SCIPI defines the pain characteristics of individuals and performs comparative analyses with clinical diagnoses. The validity and reliability properties of SCIPI were evaluated in a preliminary validation study. In this study, the following findings were obtained as a result of comparing the SCIPI with clinical diagnoses: sensitivity: 78%, specificity: 73%, and overall diagnostic accuracy: 76%. It shows that SCIPI is a reliable tool for screening neuropathic pain in individuals with spinal cord injury.
DN4 Questionnaire | 1 week
  DN4 is a questionnaire developed as a diagnostic tool that can be helpful both in daily practice and in clinical studies. It consists of 4 questions and a total of 10 items, including questions related to sensory complaints and bedside sensory examination findings, applied by the clinician. The first 2 questions are answered according to the patient's complaints, and the last 2 questions are answered according to the examination. The answers to the questions have 2 options as yes and no. Each positive item is given 1 point, and each negative item is given 0 points. The total score is calculated as the sum of 10 items, and the threshold value for neuropathic pain is determined as 4 points.
Visual Analog Scale | 1 week
  It is the most commonly used parameter to measure pain intensity. It is a self-reported scale consisting of a horizontal or vertical line, usually 10 cm long, with two verbal descriptors indicating the pain level fixed at the end points. The patient is asked to mark the point that best expresses their pain. The VAS value is obtained by considering the cm equivalent of the point they mark. '0' means no pain, '10' means unbearable pain.